Sponsor : **PROTEOR** 

## Official title:

## **Evaluation of a New Microprocessor-Controlled Prosthetic Knee :**A Prospective, Multicentered, Randomized Cross-over Trial

Unique Protocol ID: **2022-A01266-37** 

Document date: August 16, 2023

Information date: April 11, 2023

## STATISTICAL ANALYSIS PLAN

The number of participants for whom the outcome measure ware measured will be analyzed. The number of participants analyzed will be described. Expected number: 18. The population will be described in terms of anthropometric data and assigned arm.

Each subject will be included in one of 2 arms:

- Start using current MPK for 4 weeks before fitting new MPK and use it for 4 weeks OR
- Start using MPK\_NEW for 4 weeks before fitting back current MPK and use it for 4 weeks

The average PSFS score will be described for each subject and for each Microprocessor-controlled knee: current (MPK\_HAB) and new (MPK\_NEW). The main criteria measure will be **the difference of the averages** paired by the two conditions (MPK\_NEW – MPK\_HAB).

Distribution normality will be tested with Shapiro-Wilk tests; superiority tests will be run. A **t-Test, 1-sided** (student test) will be used if the dataset follows a normal distribution. Otherwise, the **Wilcoxon test** will be used. The P-value for significance is 0.05.

PSFS scores for each condition (MPK\_HAB and MPK\_NEW) will also be presented as means and standard deviations.

Secondary outcomes measures such as functional tests will be described for each condition as means and standard deviations. The t-test will be used for analysis if dataset follows a normal distribution. Otherwise, the Wilcoxon test will be used. For questionnaires, answers and scores will be analyzed for each condition.